CLINICAL TRIAL: NCT01021592
Title: Evaluation of Improvement of Quality of Life in Multiple Myeloma Patients Treated With Velcade (Bortezomib) IV: Prospective, Multicenter, Observational Study
Brief Title: Quality of Life in Multiple Myeloma Patients Treated With Bortezomib
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR012961; BOR-KOR-11
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Myeloma
Keywords: Velcade; QoL; Proteasome inhibitor; Bortezomib; EORTC QLQ C30; EQ 5D
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Injection into a vein 1.3 mg/m2 twice a week for 21 days

SUMMARY:
This observational study will observe the degree of the quality of life in patients with multiple myeloma before and after bortezomib administration by using EORTC-QLQ C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core30) and EQ-5D (EuroQol-5 Dimensions). Both tools are validated research instruments used to measure the quality of life in cancer patients and consequently will provide fundamental data regarding the quality of life in patients with multiple myeloma by analyzing factors that affect the quality of life.

DETAILED DESCRIPTION:
Many clinical studies for the treatment of multiple myeloma have been conducted in Korea, but none of them have evaluated the improvement in the quality of life in patients with multiple myeloma. Most study variables used to evaluate the quality of life of patients with multiple myeloma are subjective and limited. This study will observe the degree of change in the quality of life in patients with multiple myeloma before and after bortezomib administration by using EORTC-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core30) and EQ-5D (EuroQol-5 Dimensions), validated research instruments used to measure the quality of life in cancer patients and consequently will provide fundamental data regarding the quality of life in patients with multiple myeloma.. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients who are newly prescribed bortezomib injection as a secondary agent for the treatment of multiple myeloma
* Patients who can understand and fill out quality of life questionnaires, and who agree to provide information will be included

Exclusion Criteria:

* Patients who are hypersensitive to the bortezomib or any component of bortezomib or with a history of the hypersensitivity
* Patients with severe hepatic impairment
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients who are newly prescribed bortezomib injection as a secondary agent for the treatment of multiple myeloma, those of whom can understand and fill out questionnaire, and agree to provide information will be included.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The change in the quality of life as measured by EORTC QLQ-C30 and EQ-5D before and after the administration of bortezomib | Before the first, after the fourth and at the last IV cycle of bortezomib

SECONDARY OUTCOMES:
Relationship between the primary outcome and the complete remission (CR) rate | Before the first, after the fourth and at the last IV cycle of bortezomib
Relationship between the primary outcome and the overall response rate | Before the first, after the fourth and at the last IV cycle of bortezomib
Relationship between the primary outcome and the time to response | Before the first, after the fourth and at the last IV cycle of bortezomib
Adverse events | Every 3 week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

REFERENCES:
- See also: Evaluation in Improvement of Quality of Life in Patients with Multiple Myeloma Using Velcade® (bortezomib) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=312&filename=CR012961_CSR.pdf